CLINICAL TRIAL: NCT07352540
Title: Effects and Safety of Single Versus Triple Hyaluronic Acid Injections in the Treatment of Knee Osteoarthritis
Brief Title: Single vs Triple Hyaluronic Acid in Knee Osteoarthritis
Acronym: DR-HAKOA
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-275_1-Bm
Record Dates: First submitted 2026-01-02; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; Hyaluronic-acid; injection; safety; feasibility
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three intra-articular HA injections (Active Comparator): Three intra-articular injections of Innoryos 2.2% (2 ml each) in the knee joint at weekly intervals
  Interventions: Drug: Three intra-articular hyaluronic acid (HA) injections
- One intra-articular HA injection (Experimental): One intra-articular injection of Innoryos 2.5% (4.8 ml) in the knee joint
  Interventions: Drug: One intra-articular hyaluronic acid (HA) injection

INTERVENTIONS:
Drug: Three intra-articular hyaluronic acid (HA) injections — Therapy with intra-articular injections of hyaluronic acid (HA). Three intra-articular injections of Innoryos 2.2% (2 ml per injection) administered into the affected knee joint at weekly intervals.
  Arms: Three intra-articular HA injections
Drug: One intra-articular hyaluronic acid (HA) injection — Therapy with a single intra-articular injection of hyaluronic acid (HA). One intra-articular injection of Innoryos 2.5% (4.8 ml per injection) administered into the affected knee joint at weekly intervals.
  Arms: One intra-articular HA injection

SUMMARY:
The goal of this clinical trial is to directly compare two hyaluronic acid injection protocols in adults with knee osteoarthritis: a single intra-articular injection of Innoryos 2.5% (Single-Shot) and a three-week injection series of Innoryos 2.2% (Triple-Shot). The study aims to determine whether the single injection provides comparable safety, pain relief, and improvement in knee function to the triple-injection protocol.

The main questions are:

* How do the single-shot and triple-shot protocols compare in terms of pain reduction and functional improvement?
* How do their safety and tolerability profiles compare?
* What medical problems occur with each protocol? Participants (n = 46) will receive either the single 4.8 ml injection or three weekly 2 ml injections. They will attend clinic visits at baseline, Week 6, Week 12, and Week 24 for assessments including WOMAC score, 7-day pain diary, functional and strength tests, and MRI scans of the knee.

This single-center, partially blinded, randomized study will provide a direct comparison of the two HA injection protocols, assessing whether the single-shot approach is as safe and effective as the triple-shot regimen, while potentially offering a more convenient, patient-friendly treatment.

DETAILED DESCRIPTION:
Background:

Knee osteoarthritis (gonarthrosis) is a prevalent degenerative joint disease characterized by cartilage loss, joint pain, stiffness, and functional impairment, which significantly affects mobility and quality of life. Intra-articular injections of hyaluronic acid (HA) are a well-established conservative therapy to reduce pain, improve function, and potentially delay surgical interventions. Various HA formulations and injection protocols exist, differing in molecular weight, concentration, and dosing schedules. Optimizing treatment in terms of efficacy, safety, patient convenience, and cost-effectiveness remains a key clinical goal.

Objective:

This study aims to compare the safety, tolerability, and efficacy of a single intra-articular injection of Innoryos 2.5% (Single-Shot) with a standard three-week injection regimen of Innoryos 2.2% (Triple-Shot) in adults with moderate to severe knee osteoarthritis. The primary focus is on safety and pain reduction, with secondary outcomes including functional improvement, leg muscle strength, and structural assessment of the knee joint via MRI.

Study Design:

This is a single-center, randomized, partially blinded, parallel-group clinical intervention study including 46 participants. Patients are randomized using block randomization stratified by baseline WOMAC total score to ensure balanced distribution of baseline pain and functional impairment. Patients and treating physicians are aware of treatment allocation, while all personnel performing functional tests, MRI assessments, data entry, and statistical analyses are blinded to minimize bias.

Participants:

Adults aged 40-70 years with radiographically confirmed moderate to severe knee osteoarthritis, experiencing knee pain for at least three months and on at least 50% of days in the prior month. Key exclusion criteria include grade 4 osteoarthritis, non-osteoarthritic knee pain, other rheumatic diseases, recent HA or corticosteroid injections, recent trauma or surgery, coagulopathies, autoimmune disorders, pregnancy or lactation, and contraindications for MRI.

Interventions:

* Single-Shot Group: One intra-articular injection of Innoryos 2.5% (4.8 ml)
* Triple-Shot Group: Three intra-articular injections of Innoryos 2.2% (2 ml each) at weekly intervals

Outcomes:

The primary outcome is total WOMAC score. Secondary outcomes include WOMAC subscales, VAS pain diary, functional performance, leg muscle strength, MRI-detected structural changes, and safety/tolerability parameters.

Assessments:

Participants are assessed at baseline, Week 6, Week 12, and Week 24.

* WOMAC questionnaire (baseline, Week 6, Week 12, and Week 24): Pain, stiffness, and functional limitation
* Pain diary (VAS) (baseline, Week 6, Week 12, and Week 24): Daily for 7 days at each assessment (~1 min/day)
* Functional and strength tests (baseline, Week 6, Week 12): Chair Stand Test, Timed Up and Go Test, isokinetic leg press (~30 min per session)
* MRI (baseline, Week 6, Week 12): Baseline and Week 12 for structural assessment (~90 min including functional tests)
* Safety monitoring: Adverse events, medication use, compliance, drop-outs

Significance:

This study provides high-quality evidence for the direct comparison of single-shot versus triple-shot HA injection protocols in knee osteoarthritis. By using stratified randomization based on baseline WOMAC total score and blinded assessment of outcomes, the trial ensures unbiased evaluation. Demonstration of comparable safety and efficacy of the single-shot regimen could offer a more convenient, patient-friendly, and potentially safer therapeutic option, optimizing conservative management for patients with knee osteoarthritis.

intra-articular injection of Innoryos 2.5% (Single-Shot) with a standard three-week injection regimen of Innoryos 2.2% (Triple-Shot) in adults with moderate to severe knee osteoarthritis. The primary focus is on safety and pain reduction, with secondary outcomes including functional improvement, leg muscle strength, and structural assessment of the knee joint via MRI.

Study Design:

This is a single-center, randomized, partially blinded, parallel-group clinical intervention study including 46 participants. Patients are randomized using block randomization stratified by baseline WOMAC total score to ensure balanced distribution of baseline pain and functional impairment. Patients and treating physicians are aware of treatment allocation, while all personnel performing functional tests, MRI assessments, data entry, and statistical analyses are blinded to minimize bias.

Participants:

Adults aged 40-70 years with radiographically confirmed moderate to severe knee osteoarthritis, experiencing knee pain for at least three months and on at least 50% of days in the prior month. Key exclusion criteria include grade 4 osteoarthritis, non-osteoarthritic knee pain, other rheumatic diseases, recent HA or corticosteroid injections, recent trauma or surgery, coagulopathies, autoimmune disorders, pregnancy or lactation, and contraindications for MRI.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40-70 years
* Radiographically confirmed moderate to severe knee osteoarthritis
* Knee pain for ≥3 months
* Pain on ≥50% of days in past 30 days
* Able to provide informed consent

Exclusion Criteria:

* Grade 4 osteoarthritis (full-thickness cartilage loss)
* Non-osteoarthritic knee pain
* Other rheumatic diseases (e.g., rheumatoid arthritis, fibromyalgia)
* HA injection <6 months or corticosteroid injection <3 months in target knee
* Recent trauma or surgery of affected knee (<6 months)
* Coagulopathy or bleeding disorder
* Autoimmune or relevant systemic disease
* Dermatologic infection at injection site
* Pregnancy or lactation
* Opioid or oral corticosteroid use
* Contraindications to MRI (pacemaker, intracorporeal metal, claustrophobia)
* Expected absence during study period or noncompliance

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
WOMAC questionnaire total score | At baseline, at 6 weeks, at 12 weeks, at 24 weeks
  Total score of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), assessing overall pain, stiffness, and physical function of the knee joint

SECONDARY OUTCOMES:
WOMAC questionnaire pain subscore | At baseline, at 6 weeks, at 12 weeks, at 24 weeks
  Pain subscore of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), assessing pain of the knee joint
WOMAC questionnaire stiffness subscore | At baseline, at 6 weeks, at 12 weeks, at 24 weeks
  Stiffness subscore of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), assessing stiffness of the knee joint
WOMAC questionnaire physical function subscore | At baseline, at 6 weeks, at 12 weeks, at 24 weeks
  Physical function subscore of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), assessing pain of the knee joint
7-day pain assessment using visual analog scale (VAS) | At baseline, at 6 weeks, at 12 weeks, at 24 weeks
  Participants will record their knee pain daily using a Visual Analog Scale (VAS) as part of a 7-day pain diary at each assessment period. The VAS is a straight 100 mm line, anchored by "no pain" at 0 mm and "worst imaginable pain" at 100 mm. Participants indicate their current knee pain intensity each day by marking a point on the line that best represents their pain.
  The diary is completed for seven consecutive days to capture fluctuations in pain intensity during daily activities. The daily VAS scores are recorded and later averaged to calculate a weekly mean pain score.
Maximum isokinetic leg extension strength | At baseline, at 6 weeks, at 12 weeks, at 24 weeks
  Participants' leg muscle strength and functional performance are assessed using an isokinetic leg press (Physiomed, Laipersdorf, Germany). Before testing, participants complete a 5-minute warm-up on a cross-trainer to prepare the muscles and reduce injury risk.
  Following the warm-up, two maximal test sessions are conducted, each consisting of 6 repetitions at a velocity of 0.6 meters per second (m/s). During each attempt, participants perform the leg press extension movement with maximal effort. The highest peak force achieved during the extension in each session is recorded and used for analysis.
30-Second Chair Stand Test (30s CST) - Assessment of Lower Limb Function: | At baseline, at 6 weeks, at 12 weeks, at 24 weeks
  The 30-Second Chair Stand Test measures lower body strength, endurance, and functional mobility. Participants sit on a standard chair with arms crossed over the chest. When instructed, they stand up fully and sit back down repeatedly for 30 seconds.
  The total number of full stands completed within 30 seconds is recorded. A higher number of repetitions indicates better lower limb strength and functional performance.
Knee MRI and T2 Mapping - Assessment of Joint Structures | At baseline, at 12 weeks, at 24 weeks
  Magnetic Resonance Imaging (MRI) is used to assess structural changes in the knee joint and evaluate the integrity of cartilage and other joint tissues. Participants undergo a non-invasive, radiation-free MRI scan of the affected knee at baseline and 12 weeks after treatment.
  The MRI protocol includes high-resolution imaging of joint structures, such as cartilage, menisci, ligaments, and subchondral bone. Additionally, T2 mapping is performed to quantify the T2 relaxation time of articular cartilage, which reflects the water content and collagen organization. Areas of increased T2 values indicate cartilage degeneration or changes in cartilage composition, while decreases or stabilization suggest maintenance or improvement of cartilage health.

OTHER OUTCOMES:
Compliance and Drop-Out | up to 24 weeks
  Compliance refers to the degree to which participants adhere to the assigned injection protocol and scheduled study visits. For the Single-Shot group, compliance is assessed by confirming that participants receive the planned single 4.8 ml injection at baseline. For the Triple-Shot group, compliance is assessed by verifying that participants receive all three weekly 2 ml injections according to the study schedule. Compliance is documented in the study records and serves as a measure of treatment adherence and feasibility of the respective protocols.
  Drop-Out refers to participants who withdraw from the study before completion or fail to attend follow-up assessments at the scheduled time points (baseline, Week 6, Week 12, Week 24). Reasons for drop-out, including adverse events, personal choice, or loss to follow-up, are recorded. Drop-out rates are analyzed as an endpoint to evaluate the acceptability, tolerability, and practicality of each
Medication Use - Analgesic Tracking | Up to 24 weeks
  Participants record their use of pain medications during the 7-day pain diary period, which accompanies the daily Numeric Rating Scale (NRS) for knee pain. Each day, participants document:
  The type of pain medication taken The dosage The timing of administration
Adverse Effects - Safety Endpoint | Up to 24 weeks
  Adverse effects are monitored to assess the safety and tolerability of the hyaluronic acid injection protocols. Participants are instructed to report any adverse events or reactions following the injections. Specifically:
  Short-term monitoring: Participants record any adverse effects daily for 7 days after each injection. This includes local reactions at the injection site (e.g., pain, swelling, redness) as well as any systemic symptoms (e.g., fatigue, fever).
  Long-term monitoring: Adverse effects are also tracked throughout the entire study duration.
  All reported adverse events are documented, classified, and analyzed according to severity, duration, and possible relation to the treatment.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared publicly in order to comply with data protection regulations in Germany (GDPR) and the study's data protection consent. Only aggregated and anonymized results will be reported in publications or study summaries. No personal identifiers, contact information, or sensitive participant data will be disclosed.

REFERENCES:
- [Background] Kast S, Kemmler W, Roemer FW, Kohl M, Culvenor AG, Mobasheri A, Uder M, von Stengel S. Effectiveness of whole-body electromyostimulation on knee pain and physical function in knee osteoarthritis: a randomized controlled trial. Sci Rep. 2024 Sep 6;14(1):20804. doi: 10.1038/s41598-024-71552-7. PMID 39242729
- [Background] Roemer FW, Kast S, Kemmler W, Collins JE, Engelke K, Guermazi A, Uder M, von Stengel S. Structural effects of whole body electromyostimulation on knee osteoarthritis: the EMSOAT Study. Skeletal Radiol. 2025 Nov;54(11):2579-2588. doi: 10.1007/s00256-025-04984-5. Epub 2025 Jul 22. PMID 40694090
- [Background] Hofweber, L., von Stengel, S., Nürnberger, J., & Kemmler, W. (2024). Effectiveness and safety of the hyaluronic acid INNORYOS 2.2% in patients with early to advanced knee osteoarthritis. A prospective non-interventional randomized clinical trial.